## Patient Education to Improve Pain Management in Older Adults with Acute Musculoskeletal Pain: A Pilot Randomized Trial

**Statistical Analysis Plan** 

NCT02438384

July 25, 2015

Descriptive statistics will be used to present baseline characteristics for patients in each of the three study arms. To characterize the primary outcome by intervention arm, we will calculate point estimates along with 95% confidence intervals for change in average pain scores from baseline to one month with adjustments made for age, gender, and baseline pain scores. Pairwise difference in change in average pain between each of the three possible comparison pairs (video plus telecare vs. usual care, video alone vs. usual care, video plus telecare vs. video alone) will also be estimated along with 95% confidence intervals, adjusted for baseline pain, age and gender. Process outcomes will also be described using descriptive statistics.